CLINICAL TRIAL: NCT00573534
Title: Pilot Study of Vyvanse™ (Lisdexamfetamine Dimesylate) in Adolescents (Ages 11-15) With ADHD and an Older Sibling With ADHD and Substance Dependence
Brief Title: Pilot Study of Vyvanse™ In ADHD Adolescents at Risk for Substance Abuse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5522
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2011-11-29 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2016-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; ADD; Prevention; Substance use; Adolescent
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Vyvanse (Experimental): Open Label Vyvanse (lisdexamphetamine) in doses of 30-70 mgs over 8 weeks in younger siblings of substance abusing older siblings with a history of treatment for ADHD
  Interventions: Drug: Vyvanse

INTERVENTIONS:
Drug: Vyvanse — Patients will be titrated from 30 mgs to 50 mgs to 70 mgs over four weeks, as tolerated and as needed to control ADHD symptoms
  Other Names: Lisdexamphetamine is marketed as Vyvanse

SUMMARY:
This is an open label pilot study to obtain information on the best way to study young adolescents with Attention Deficit Hyperactivity Disorder (ADHD)who may also be at risk of developing substance abuse, in part because of their ADHD. The plan is to recruit older children/young adolescents (age 11-15) who have ADHD and also have an older sibling with substance abuse. The treatment for ADHD in the 11-15 year old will be Vyvanse, a novel preparation of dextroamphetamine in which the molecule is inactivated and only becomes activated when it is digested. This preparation is felt to be safer from diversion while at the same time providing treatment for the younger siblings in which a bad outcome has already occurred in the family, namely the older sibling's substance abuse. As mentioned, this is an open-label study, a feasibility study to see if we can use this approach to study and treat high risk youth before they develop substance abuse.

DETAILED DESCRIPTION:
The study is a six month open-label treatment with Vyvanse, a novel preparation of the Attention Deficit Hyperactivity Disorder (ADHD) medication dextroamphetamine in which the drug is inactivated and only becomes reactivated when digested. Vyvanse is thought to be safer in youth at risk for substance use disorder because it is harder to abuse and divert. It is FDA approved to treat ADHD in children age 6 through 12. Although there are no negative studies in adolescents 13-15, efficacy has not been established in the latter age group.

In this study 30 adolescents (ages 11-15) will be identified who have Attention Deficit Disorder and are at risk for alcohol and substance use problems. We propose to treat their Attention Deficit Hyperactivity Disorder with Vyvanse in the hope that it may prevent ADHD from promoting the development of alcohol and substance abuse problems. Our main goal is to see if we can identify children who are at risk because they have an older sibling who already has a substance abuse problem and Attention Deficit Hyperactivity Disorder. This is dubbed "the younger sibling design." Families will be recruited via contacts in adolescent substance abuse treatment centers (e.g. Phoenix House, Odyssey House). Participating substance abuse treatment centers will inform families of our study. We will conduct two phone screens followed by an in person evaluation to determine eligibility. Relevant information includes family history with special emphasis on the growth and development of both children, as well as the results of a comprehensive clinical evaluation of the younger child. Subjects will therefore be the younger siblings of substance abusers in which both sibs have ADHD but only the older sib uses drugs or alcohol regularly. All subjects will receive active medication and all will be assessed weekly for the first three months of the study and monthly for three months thereafter. The assessments will focus on ADHD symptoms, substance use, and overall adolescent problem behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV-TR criteria for ADHD
* Has a Gender-Matched older sibling with ADHD and substance dependence
* Medically healthy
* Parents give informed consent
* Child gives assent

Exclusion Criteria:

* Significant use of alcohol or marijuana (more than ten episodes) in the past 30 days or any use of cocaine or opiates in the past 30 days; significant nicotine use is not an exclusion
* History of cardiac abnormality, past cardiac problems or family history of the same, history of fainting, open-heart surgery, and arrhythmia
* History of paranoia on stimulant medication
* Seizure or other neurological disturbance
* Pregnancy
* Moderate to severe mental deficiency as determined by IQ <60 or placement in special education for mental deficiency
* Physical exam or laboratory results with significant abnormalities
* Active suicidal or homicidal ideation or history of suicide attempts
* Unequivocal manic or hypomanic episode
* Sexually active females who are unwilling to use effective methods of contraception
* Psychosis or psychosis in a first degree relative
* Current Major Depression
* Individuals who have previously seen a cardiologist until reevaluated by a cardiologist
* Individuals for whom the current cardiac evaluation is not definitive until seen by a cardiologist and given an echocardiogram
* Individuals with Tic disorder
* Significant co-morbid anxiety disorders (i.e., OCD, Panic, PTSD)
* ADHD in remission on another psychostimulant or not in remission but in the context of inadequate dosing of a currently prescribed and administered other psychostimulant

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Donovan, MD, Principal Investigator — Columbia University / New York State Psychiatric Institute

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from March 2008 until January 2010 from parents with adolescent children in adolescent substance use treatment center and with parents of children with ADHD whether there were older children who might have substance use problems. Community pediatricians and child psychiatrists supplemented this approach.
Pre-assignment Details: This was an open-label study, hence no group assignment. Thirteen families were offered study participation, 8 accepted. The five families that declined participation cited the impracticality of weekly visits and/or the adolescent's oppositional behavior as primary reasons for nonparticipation.
Groups:
- Group 1: Adolescents with ADHD and an older sibling with Substance Use Disorder
Period: Overall Study
Arm/Group | Group 1
Started | 8
Completed | 5
Not Completed | 3
Not completed — oppositional behavior | 3

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (2)
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 70% Reduction in ADHD Symptoms as Measured by Change in ADHD Rating Scale From First to Last Visit
Description: The outcome is the number of subjects who achieved a clinically meaningful reduction in ADHD symptoms. This is defined as a 70% reduction from baseline as measured by change in the ADHD Rating Scale (ADHD-RS). The ADHD RS quantifies symptoms on a 0-3 scale, 0 meaning never present, 1 sometimes, 2 often present, 3 very often present. For this study, the scale was clinician administered using both parent and adolescent to achieve a consensus score, or a best estimate on the clinician's part when consensus could not be achieved
Time Frame: up to 24 weeks
Population: All patients who agreed to participate. Last Observation Carried Forward was used final outcome.
Measure: Number; unit: participants
Groups:
- Group 1: Lisdexamfetamine and family counseling
Arm/Group | Group 1
Number analyzed (Participants) | 8
participants
  much improved (70 percent or more drop in ADHD-RS) | 6 (0)
  unimproved | 2 (0)

2. Secondary Outcome: Number of Participants With Low or no Substance Use During the Study vs the Number With Intermittent Use Judged by (1)Time Line Follow Back (Confidential Clinician Administered Record of Recent Substance Use) (2) Urine Toxicology.
Description: This outcome measure integrates data from self report supplied in the Time Line Follow Back (a self report summary of all substance and alcohol use over the previous week or month) with evidence from periodic (weekly to monthly) urine toxicologies.
Time Frame: up to 24 weeks
Population: The 8 subjects who took at least one dose of the medication and returned for follow up were included.
Measure: Number; unit: participants
Groups:
- Lisdexamfetamine Plus Family Therapy: patients received lisdexamfetamine up to 70 mgs plus family counseling
Arm/Group | Lisdexamfetamine Plus Family Therapy
Number analyzed (Participants) | 8
participants
  none-low | 5 (0)
  intermittent | 3 (0)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected over 20 months.
Groups:
- Group 1: Intervention with Vyvanse
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No